CLINICAL TRIAL: NCT00241904
Title: Reducing Total Cardiovascular Risk in an Urban Community
Acronym: COACH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 335; R01HL082638 (NIH); NCT00385619 (obsolete NCT alias)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Diabetes Mellitus; Atherosclerosis; Cerebral Arteriosclerosis; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Diabetes Mellitus; Atherosclerosis; Intracranial Arteriosclerosis; Hypertension | interventions — Platelet Aggregation Inhibitors; Aspirin; Adrenergic beta-Antagonists; Metoprolol; Atenolol; Propranolol; Angiotensin-Converting Enzyme Inhibitors; Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Comprehensive Intervention Group (Active Comparator): The NP/CHW intervention focused on behavioral interventions to affect therapeutic lifestyle changes and adherence to medications and appointments as well as the prescription and titration of medications for one year. The NP and CHW worked as a team. The NP oversaw the initial assessment and, in collaboration with the CHW, tailored the intervention plan, conducted the intervention including lifestyle modification counseling and medication titration and prescription, consulted with the physician, and supervised the CHW. Specific algorithms for drug treatment of hyperlipidemia, hypertension (HBP), hyperglycemia, ACE, and β-blocker therapy were developed for this study based on current guidelines and standards of care.
  Interventions: Behavioral: Lifestyle Changes; Drug: Antiplatelet Agents; Drug: Beta Blocker; Drug: ACE Inhibitors
- Less Intensive Intervention Group (Active Comparator): Participants will receive usual care from their physicians and a Less Intensive (LI) intervention of feedback on cardiovascular disease (CVD) risk factors and guidelines to patients and their physicians. Patients and their providers in the received the results of baseline lipids, BP, and HbA1c along with the recommended goal levels and a pamphlet on controlling risk factors published by the American Heart Association. In addition, providers received copies of the AHA/ACC Guidelines for Secondary Prevention.
  Interventions: Behavioral: Lifestyle Changes

INTERVENTIONS:
Behavioral: Lifestyle Changes — Nutrition counseling, smoking cessation counseling, medication compliance counseling, exercise
Drug: Antiplatelet Agents — Aspirin 81 mg q day
  Other Names: Bayer, Ecotrin
  Arms: Comprehensive Intervention Group
Drug: Beta Blocker — Oral medication
  Other Names: Metoprolol; Toprol; Atenolol; Propranolol
  Arms: Comprehensive Intervention Group
Drug: ACE Inhibitors — Oral medications, received 1-2 times per day
  Other Names: Lisinopril
  Arms: Comprehensive Intervention Group

SUMMARY:
PLEASE NOTE: THIS STUDY IS ONLY ENROLLING PATIENTS CURRENTLY BEING TREATED AT BELAIR-EDISON FAMILY HEALTH CENTER.

The purpose of this study is to compare the clinical effectiveness and cost effectiveness of two cardiovascular risk reduction programs - a comprehensive intensive (Cl) intervention with a less intensive (LI) intervention - in African American, and white low-income patients with known excessive cardiovascular disease risk.

DETAILED DESCRIPTION:
BACKGROUND:

The study is based on the premise that a community-based participatory research partnership model, using a team of an advanced practice nurse case manager, community health worker (CHW), and physician can be translated into urban community clinics and improve the quality of care and reduce disparities in cardiovascular health in minority and other underserved populations. Despite well-publicized guidelines on the appropriate management of cardiovascular disease (CVD) and type 2 diabetes, implementation of CVD risk-reducing practices remains poor. In spite of the known benefit of lowering low-density lipoprotein cholesterol (LDL-C) levels below 100 mg/dl in persons with existing heart disease, as many as 50 to 70 percent of eligible CVD patients are not placed on lipid-lowering therapy by their providers and from 20 to 80 percent of patients do not achieve the goals of therapy. The benefits of controlling high blood pressure (HBP) are well established, yet national rates of HBP control remain at only 31 percent despite decades of provider and patient education. In addition, it is well established that control of glycemia, hyperlipidemia, and blood pressure reduce the risk of vascular complications in people with diabetes, 75 percent of whom die from some form of heart or blood vessel disease. This randomized trial will compare the clinical effectiveness and cost effectiveness of a CI intervention with a LI intervention in African American, and white low-income patients with known excessive CVD risk.

DESIGN NARRATIVE:

Eligible patients with CVD or type 2 diabetes will be randomly selected from two urban federally funded community clinics and randomly assigned to receive either 1) a Cl intervention delivered by a nurse practitioner, a CHW, and the patient's physician, focusing on behavioral interventions to affect therapeutic lifestyle changes and medication adherence as well as the prescription and titration of medications or 2) a LI intervention providing feedback on CVD risk factors and guidelines to patients and their physicians. Outcomes will be measured at baseline and one and two years. It is hypothesized that a higher proportion of patients in the Cl intervention group will achieve the treatment goals for lipid, blood pressure, and diabetes management, lifestyle behaviors and utilization of antiplatelet agent, beta blocker, and angiotensin converting enzyme (ACE) inhibitor therapies and that the Cl intervention will be cost-effective. Secondary outcomes include assessment of the impact of the Cl intervention model on patients' satisfaction with care and health care utilization. The increase in the percentage of high-risk women and men who receive recommended secondary prevention therapies and achieve goal levels could potentially result in a marked decrement in annual CVD mortality and health disparities if applied within primary care settings to populations with the characteristics of the target groups for this study.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving medical care at Johns Hopkins University
* African American or Caucasian and have diagnosed CVD, defined as a prior myocardial infarction, revascularization procedure for coronary disease, ischemic heart disease, stroke, or have diagnosed type 2 diabetes and not receiving any therapy
* Have either no LDL-C in their medical record during the 12 months prior to study entry or have an LDL greater than or equal to 100 mg/dl on or off lipid lowering pharmacotherapy
* Have either no blood pressure recorded in their medical record during the 12 months prior to study entry or a BP greater than 140/90 mmHg or greater than 130/80 mmHg if the participant is diabetic or has renal insufficiency
* If the participant is diabetic he or she has to either have no HbA1c recorded during the 12 months prior to study entry or HbA1c of 7 percent or greater

Exclusion criteria:

* A serious life-threatening noncardiac comorbidity with a life expectancy of less than 5 years
* A serious physician-recorded psychiatric morbidity that would interfere with the study
* Sufficient neurological impairment that would interfere with the study

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2006-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerilyn Allen, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Researchers can contact the PI for access to the data set

REFERENCES:
- [Derived] Allen JK, Dennison-Himmelfarb CR, Szanton SL, Bone L, Hill MN, Levine DM, West M, Barlow A, Lewis-Boyer L, Donnelly-Strozzo M, Curtis C, Anderson K. Community Outreach and Cardiovascular Health (COACH) Trial: a randomized, controlled trial of nurse practitioner/community health worker cardiovascular disease risk reduction in urban community health centers. Circ Cardiovasc Qual Outcomes. 2011 Nov 1;4(6):595-602. doi: 10.1161/CIRCOUTCOMES.111.961573. Epub 2011 Sep 27. PMID 21953407

RESULTS

PARTICIPANT FLOW:
Groups:
- Comprehensive Intervention Group: Participants will receive a Comprehensive Intervention (CI) delivered by a nurse practitioner, a CHW, and the patient's physician, focusing on behavioral interventions to affect therapeutic lifestyle changes in diet, exercise and medication adherence as well as the prescription and titration of medications prescribed according to study algorithms.Participants will receive a LI intervention providing feedback on CVD risk factors and guidelines to patients and their physicians.
  Lifestyle Changes: Nutrition counseling, smoking cessation counseling, medication compliance counseling, exercise
  Antiplatelet Agents: Aspirin 81 mg q day
  Beta Blocker: Oral medication
  ACE Inhibitors: Oral medications, received 1-2 times per day
- Less Intensive Intervention (Usual Care) Group: Participants will receive usual care from their physicians and a Less Intensive (LI) intervention of feedback on cardiovascular disease (CVD) risk factors and guidelines to patients and their physicians.
Period: Overall Study
Arm/Group | Comprehensive Intervention Group | Less Intensive Intervention (Usual Care) Group
Started | 261 | 264
Completed | 227 | 240
Not Completed | 34 | 24

BASELINE CHARACTERISTICS:
Groups:
- Comprehensive Intervention: CI intervention will receive Behavioral: Lifestyle Changes, Nutrition counseling, smoking cessation counseling, medication compliance counseling, exercises, as well as pharmacologic agents
- Less Intensive Intervention: LI Arm: Participants will receive usual care from their physicians and a Less Intensive (LI) intervention of feedback on cardiovascular disease (CVD) risk factors and guidelines to patients and their physicians.
- Total: Total of all reporting groups
Arm/Group | Comprehensive Intervention | Less Intensive Intervention | Total
Number analyzed (Participants) | 261 | 264 | 525
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (12) | 54.7 (11.5) | 54.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 187 | 374
  Male | 74 | 77 | 151
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 207 | 210 | 417
  White | 54 | 54 | 108

OUTCOME MEASURES:

1. Primary Outcome: Low-density Lipoprotein Cholesterol
Description: Blood was drawn after a 12 hour fast and low density lipoprotein cholesterol was measured in a standardized lab
Time Frame: Measured at 1 year
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Comprehensive Intervention Group: Participants will receive a Comprehensive Intervention (CI) delivered by a nurse practitioner, a CHW, and the patient's physician, focusing on behavioral interventions to affect therapeutic lifestyle changes in diet, exercise and medication adherence as well as the prescription and titration of medications prescribed according to study algorithms for antiplatelet agents, beta blockers, ace inhibitors..
  Lifestyle Changes: Nutrition counseling, smoking cessation counseling, medication compliance counseling, exercise
  Antiplatelet Agents: Aspirin 81 mg q day
  Beta Blocker: Oral medication
  ACE Inhibitors: Oral medications, received 1-2 times per day
- Less Intensive Intervention Group: Participants will receive usual care from their physicians and a Less Intensive (LI) intervention of feedback on cardiovascular disease (CVD) risk factors and guidelines to patients and their physicians.
  Antiplatelet Agents: Aspirin 81 mg q day
  Beta Blocker: Oral medication
  ACE Inhibitors: Oral medications, received 1-2 times per day
Arm/Group | Comprehensive Intervention Group | Less Intensive Intervention Group
Number analyzed (Participants) | 261 | 264
mg/dL | 100.1 (39.2) | 110.6 (36.8)
Statistical Analysis 1: Comparison: Comprehensive Intervention Group vs Less Intensive Intervention Group; Intention to treat analysis was used; Test type: Superiority; p < 0.001, General Linear Mixed Model

2. Primary Outcome: Systolic Blood Pressure
Description: Blood pressure measured with automatic blood pressure machine according to the guidelines of the American Heart Association.
Time Frame: Measured at 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Comprehensive Intervention Group | Less Intensive Intervention Group
Number analyzed (Participants) | 261 | 264
mmHg | 130.8 (20.7) | 135.9 (20.5)
Statistical Analysis 1: Comparison: Comprehensive Intervention Group vs Less Intensive Intervention Group; Test type: Superiority; p = 0.003, General Linear Mixed Model

3. Primary Outcome: HbA1c
Description: Fasting for 12 hour blood sample was measured in standardized lab
Time Frame: Measured at 1 year
Population: Only the participants with a diagnosis of diabetes were assessed for this outcome measure
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Groups:
- Comprehensive Intervention Group: Participants will receive a Comprehensive Intervention (CI) delivered by a nurse practitioner, a CHW, and the patient's physician, focusing on behavioral interventions to affect therapeutic lifestyle changes in diet, exercise and medication adherence as well as the prescription and titration of medications prescribed according to study algorithms for antiplatelet agents, beta blockers, ace inhibitors..
  Lifestyle Changes: Nutrition counseling, smoking cessation counseling, medication compliance counseling, exercise
  Antiplatelet Agents: Aspirin 81 mg q day
  Beta Blocker: Oral medication
  ACE Inhibitors:Oral medications, received 1-2 times per day
Arm/Group | Comprehensive Intervention Group | Less Intensive Intervention Group
Number analyzed (Participants) | 104 | 110
percentage of hemoglobin | 8.3 (2.2) | 8.2 (2.1)
Statistical Analysis 1: Comparison: Comprehensive Intervention Group vs Less Intensive Intervention Group; Test type: Superiority; p = 0.034, General Linear Mixed Model

4. Secondary Outcome: Patients' Satisfaction With Care and Health Care Utilization
Description: Patient satisfaction with care and healthcare utilization was measured with the Patient Assessment for Chronic Illness Care Scale (PACIC). The scores range from 0-5, with 5 being the most satisfied
Time Frame: Measured at 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comprehensive Intervention Group | Less Intensive Intervention Group
Number analyzed (Participants) | 261 | 264
units on a scale | 2.9 (0.9) | 1.8 (1.0)
Statistical Analysis 1: Comparison: Comprehensive Intervention Group vs Less Intensive Intervention Group; Test type: Superiority; p < 0.001, General Linear Mixed Model

ADVERSE EVENTS:
Arm/Group | Comprehensive Intervention Group | Less Intensive Intervention
Serious Adverse Events (participants affected / at risk) | 0/261 | 0/264
Other Adverse Events (participants affected / at risk) | 0/261 | 0/264

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No